CLINICAL TRIAL: NCT02316548
Title: Randomized Phase II Trial of Postoperative Adjuvant IMRT Following Cystectomy for pT3/T4 Urothelial Bladder Cancer
Brief Title: Surgery With or Without Postoperative Intensity Modulated Radiation Therapy in Treating Patients With Urothelial Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial will not meet CTEP Early Phase Trial Slow Accrual Guidelines
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU001; NCI-2014-02061 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU001 (Other: NRG Oncology); NRG-GU001 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: Stage III Bladder Cancer; Stage IV Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Radiation Therapy (No Intervention): Patients do not receive radiation therapy (RT).
- Intensity-modulated radiation therapy (IMRT) (Experimental): Postoperative adjuvant intensity-modulated radiation therapy (IMRT).
  Interventions: Radiation: Intensity-Modulated Radiation Therapy

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Postoperative adjuvant IMRT radiotherapy 50.4 Gy in 28 fractions. In patients not getting postoperative adjuvant chemotherapy the radiation treatment must begin within 140 days after cystectomy. For patients getting adjuvant chemotherapy radiation treatment must start within 49 days of completing chemotherapy.
  Other Names: IMRT
  Arms: Intensity-modulated radiation therapy (IMRT)

SUMMARY:
This randomized phase II trial studies the side effects and how well postoperative intensity modulated radiotherapy works after surgery in treating patients with urothelial bladder cancer. Radiation therapy uses high energy x-rays to kill tumor cells left behind in the pelvis after surgery. It is not yet known whether surgery followed by radiotherapy is more effective than surgery alone in treating patients with urothelial bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the ability of postcystectomy adjuvant radiotherapy to safely reduce pelvic tumor recurrence, defined as pelvic recurrence-free survival.

SECONDARY OBJECTIVES:

I. Evaluate increase in disease-free survival. II. Evaluate toxicity of adjuvant pelvic radiotherapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms. Patients are stratified by neoadjuvant preoperative or postoperative adjuvant chemotherapy.

After completion of study treatment, patients are followed up at 6 weeks, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria (A patient cannot be considered eligible for this study unless ALL of the following conditions are met.):

* Initial histological diagnosis of muscle invasive urothelial carcinoma
* Patients must have undergone a radical cystectomy (reconstructed urinary diversion may be non-continent diversions (eg, ileal conduits) or continent non-orthotopic catheterizable diversions (eg, Indiana pouch) or continent orthotopic diversions (eg, Studer pouch or neobladder)for urothelial bladder carcinoma within 105 days prior to registration. Final cystectomy pathology must be either pure urothelial carcinoma or dominant urothelial carcinoma with admixture of other histologies excluding small cell variants.

  * Neoadjuvant (preoperative) or adjuvant (postoperative) chemotherapy for the bladder cancer is permitted; however, all patients, even those who will receive adjuvant chemotherapy, must be registered within 105 days after completing cystectomy regardless of whether adjuvant chemotherapy has started. Patients who will be receiving adjuvant (postoperative) chemotherapy will be randomized within 28 days of completing that chemotherapy.
* Patients with the following pTNM stages per the American Joint Committee on Cancer (AJCC) 7th ed. are eligible:

  * pT3apN0; pN1; pN2 provided less than 10 nodes dissected and/or positive surgical margins
  * pT3bpN0; pN1; pN2
  * pT4apN0; pN1; pN2
  * pT4bpN0; pN1; pN2
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination =< 45 days prior to registration;
  * CT or MRI or positron emission tomography(PET)-CT that includes chest, abdomen and pelvis should be performed for initial radiological staging. This may be performed pre- or post-surgery ≤ 90 days prior to registration except in patients getting postoperative adjuvant chemotherapy, who will require CT, MRI or PET-CT including the chest and abdomen and pelvis no more than 30 days prior to registration. Imaging performed postoperatively should show no evidence of residual disease.
* Age >=18
* Zubrod performance status 0-2 =< 45 days prior to registration
* Complete blood count (CBC)/differential obtained ≤ 14 days prior to registration with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
  * Platelets >= 100,000 cells/mm^3
  * Hemoglobin >= 8.0 g/dl (NOTE: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
  * The patient must provide study-specific informed consent prior to study entry
* The patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria (Patients with any of the following conditions are NOT eligible for this study.):

* Definitive clinical or radiologic evidence of metastatic disease; pN3 disease is not allowed (positive common iliac node).
* Prior invasive solid tumor or hematological malignancy (except non-melanomatous skin cancer and incidentally discovered prostate cancer at time of cystoprostatectomy) unless disease free for a minimum of 3 years
* Prior radiotherapy to the pelvis
* Patients with a history of inflammatory bowel disease
* Patients who have required any treatment (medical or surgical) for bowel obstruction prior to diagnosis of bladder cancer or who have required surgical treatment for bowel obstruction after the cystectomy
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
  * Transmural myocardial infarction within the last 6 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Severe hepatic disease, defined as a diagnosis of Child-Pugh Class B or C hepatic disease;
  * HIV positive with CD4 count < 200 cells/microliter. Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter within 30 days prior to registration. Note also that HIV testing is not required for eligibility for this protocol.
  * Other major medical illness which requires hospitalization or precludes study therapy at the time of registration.
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Libni Eapen, Principal Investigator — NRG Oncology
Locations (127):
- United States (116):
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Marin General Hospital, Greenbrae, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Virtua Memorial, Mount Holly, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Bay Area Hospital, Coos Bay, Oregon
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (10):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Rabin Medical Center, Petah Tikva, Israel

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fourteen patient were screened. One patients did not continue to randomization due to disease progression and was not followed further.
Groups:
- Intensity-modulated Radiation Therapy (IMRT): Postoperative adjuvant IMRT radiotherapy 50.4 Gy in 28 fractions.
Period: Overall Study
Arm/Group | No Radiation Therapy | Intensity-modulated Radiation Therapy (IMRT)
Started | 6 (Randomized) | 7 (Randomized)
Eligible Population | 6 | 6
Eligible With Disease Assessment | 4 | 1
Eligible With Adverse Event Data | 4 | 2
Completed | 6 (Eligible patients on study until study termination) | 6 (Eligible patients on study until study termination)
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | No Radiation Therapy | Intensity-modulated Radiation Therapy (IMRT) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Full Range); unit: years] | 67 [60 to 77] | 67 [37 to 82] | 67 [37 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Chemotherapy [Count of Participants; unit: Participants]
  Neoadjuvant or adjuvant chemotherapy | 5 | 4 | 9
  No chemotherapy | 1 | 2 | 3
Pelvic Relapse Risk Category [Count of Participants; unit: Participants] — Intermediate risk= pT3b/pT4a/pT4b pN0-2 with negative margins and 10 or more nodes dissected. High risk = pT3a/pT3b/pT4a/pT4b pN0-2 with less than 10 nodes dissected and/or with positive margins.
  Participants
    Intermediate Risk | 3 | 3 | 6
    High Risk | 3 | 3 | 6
Zubrod performance status [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 2 | 3 | 5
    1 | 2 | 3 | 5
    2 | 2 | 0 | 2
T Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 7th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T3a | 2 | 0 | 2
    T3b | 3 | 2 | 5
    T4a | 1 | 3 | 4
    T4b | 0 | 1 | 1
N Stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per the AJCC 7th ed. refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    N0 | 3 | 2 | 5
    N1 | 2 | 3 | 5
    N2 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Recurrence-free Survival (PRFS)
Description: PRFS is defined as time free of pelvic recurrence or death, with patients who experience distant metastasis censored at the time of occurrence. Pelvic recurrence is specifically defined as soft tissue and /or lymph node tumor recurrence in the pelvis anywhere between the L5-S1 disc space superiorly and the pelvic floor inferiorly. This was to be determined on the basis of pelvic imaging (CT or MRI scan demonstrating soft tissue or nodal recurrence at least 1cm in linear dimension) or urethroscopy; biopsy was not required. PRFS was to be tested between arms in terms of a difference in cause-specific-hazards using the log-rank test and cumulative incidence of PRFS in the presence of competing risks was to be computed via cumulative incidence. Due to early termination with few patients, only counts of events have been calculated.
Time Frame: From randomization to study termination, maximum follow-up was 13.3 months, median follow-up was 1.9 months
Population: Randomized eligible patients with disease assessment data
Measure: Count of Participants; unit: Participants
Arm/Group | No Radiation Therapy | Intensity-modulated Radiation Therapy (IMRT)
Number analyzed (Participants) | 4 | 1
Participants | 1 | 0

2. Secondary Outcome: Disease Free Survival (DFS)
Description: Disease free survival (DFS) is defined as the first occurrence of either: pelvic failure, distant metastasis, or death and was to be estimated by the Kaplan-Meier method and arms compared using the log-rank test. Pelvic recurrence is specifically defined as soft tissue and /or lymph node tumor recurrence in the pelvis anywhere between the L5-S1 disc space superiorly and the pelvic floor inferiorly. This was to be determined on the basis of pelvic imaging (CT or MRI scan demonstrating soft tissue or nodal recurrence at least 1cm in linear dimension) or urethroscopy; biopsy was not required. Distant metastases is defined as any hematogenous metastases and/or lymph node metastases above the L5-S1 interspace, documented by imaging (CT and/or MRI and/or bone scans). Due to early termination with few patients, only counts of events have been calculated.
Time Frame: From randomization to study termination, maximum follow-up was 13.3 months, median follow-up was 1.9 months
Population: Randomized eligible patients with disease assessment data
Measure: Count of Participants; unit: Participants
Arm/Group | No Radiation Therapy | Intensity-modulated Radiation Therapy (IMRT)
Number analyzed (Participants) | 4 | 1
Participants | 2 | 1

3. Secondary Outcome: Number of Patients With Bowel Toxicity
Description: Adverse events (AE) evaluated using Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Bowel toxicity= abdominal distension/pain, colitis, colonic fistula/ hemorrhage/obstruction/perforation/stenosis/ulcer, diarrhea, enterocolitis, fecal incontinence/gastrointestinal/fistula/pain, ileal fistula/hemorrhage/obstruction/perforation/stenosis/ulcer, Ileus, jejunal fistula/hemorrhage/obstruction/perforation/stenosis/ulcer, lower gastrointestinal hemorrhage, rectal fistula/hemorrhage/mucositis/necrosis/obstruction/pain/perforation/stenosis/ulcer, small intestinal mucositis/obstruction/perforation/stenosis/ulcer, vomiting. Highest grade adverse event per subject counted. Grade refers to AE severity and ranges from 1 to 5 with unique clinical descriptions of severity for each AE based on this general guideline: 1 Mild, 2 Moderate, 3 Severe, 4 Life-threatening or disabling, 5 Death related to AE.
Time Frame: From randomization to study termination, maximum follow-up was 13.3 months, median follow-up was 1.9 months
Population: Randomized eligible patients with adverse event data
Measure: Count of Participants; unit: Participants
Arm/Group | No Radiation Therapy | Intensity-modulated Radiation Therapy (IMRT)
Number analyzed (Participants) | 4 | 2
Participants
  None | 2 | 0
  Grade 1 | 2 | 1
  Grade 2 | 0 | 0
  Grade 3 | 0 | 1
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization to study termination, maximum follow-up was 13.3 months, median follow-up was 1.9 months.
Description: Randomized eligible patients with adverse event data are included in the adverse event tables. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event. All randomized eligible patients are include in the mortality table.
Arm/Group | No Radiation Therapy | Intensity-modulated Radiation Therapy (IMRT)
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/2
Other Adverse Events (participants affected / at risk) | 3/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No Radiation Therapy (N=4) | Intensity-modulated Radiation Therapy (IMRT) (N=2)
Diarrhea (Gastrointestinal disorders) | 0 | 1
Rectal fistula (Gastrointestinal disorders) | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No Radiation Therapy (N=4) | Intensity-modulated Radiation Therapy (IMRT) (N=2)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study stopped accrual early due to unmet targeted accrual goals with 14 subjects accrued out of 185 planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT02316548/Prot_SAP_000.pdf